CLINICAL TRIAL: NCT00746798
Title: Randomized, Modified, Double-blind, Placebo-controlled, Phase II, Dose-ranging Study of the Safety and Immunogenicity of Single Dose ChimeriVax-WN02 Vaccine in Healthy Adults.
Brief Title: Safety and Immunogenicity Study of ChimeriVax West Nile Vaccine in Healthy Adults
Acronym: WinVax004
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Sanofi Pasteur, a Sanofi Company (Industry)
Responsible Party: Sponsor
Organization: Sanofi (Industry)
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Prevention
Other Study IDs: H-244-004
Record Dates: First submitted 2008-09-02; First posted 2008-09-04 (Estimated); Results first posted 2011-11-02 (Estimated); Last update posted 2015-04-03 (Estimated); Status verified 2015-03

CONDITIONS: West Nile Fever
Keywords: West Nile Fever; ChimeriVax; West Nile Virus Vaccine
MeSH Terms: conditions — West Nile Fever

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (4):
- ChimeriVax WN02 vaccine, low dose (Experimental): Participants randomized to receive ChimeriVax WN02 vaccine, low dose
  Interventions: Biological: ChimeriVax-WN02 vaccine
- ChimeriVax-WN02 vaccine, medium dose (Experimental): Participants randomized to receive ChimeriVax-WN02 vaccine, medium dose
  Interventions: Biological: ChimeriVax-WN02 vaccine
- ChimeriVax-WN02 vaccine, high dose (Experimental): Participants randomized to receive ChimeriVax-WN02 vaccine, high dose
  Interventions: Biological: ChimeriVax-WN02 vaccine
- Placebo (Placebo Comparator): Participants randomized to receive Placebo (Saline)
  Interventions: Biological: Placebo

INTERVENTIONS:
Biological: ChimeriVax-WN02 vaccine — low dose, approximately 4 x 3log10, given one time subcutaneously
  Arms: ChimeriVax WN02 vaccine, low dose
Biological: ChimeriVax-WN02 vaccine — medium dose, approximately 4 x 4log10, given one time
  Arms: ChimeriVax-WN02 vaccine, medium dose
Biological: ChimeriVax-WN02 vaccine — high dose, approximately 4 x 5log10, given one time subcutaneously
  Arms: ChimeriVax-WN02 vaccine, high dose
Biological: Placebo — 0.9%Normal Saline for Injection, given one time subcutaneously
  Arms: Placebo

SUMMARY:
The purpose of this study is to determine if ChimeriVax West Nile vaccine is safe and effective in preventing West Nile disease in adults over 50 years of age.

DETAILED DESCRIPTION:
Currently, the only method of prevention of West Nile infection is control of the mosquito vectors associated or avoidance of mosquito bites, which has proven largely ineffective. Developing a safe, effective vaccine and making it widely available will enhance the prospects of prevention and control of this disease. In addition, natural infections with the YF virus and WN virus are more severe in the elderly. Therefore, a study among healthy older subjects or those with well controlled chronic diseases will provide data to determine a ChimeriVax-WN02 vaccine dose that is immunogenic and well tolerated.

ELIGIBILITY:
Inclusion Criteria:

* Written informed consent
* Medically stable, ambulatory male or female ≥ 50 years of age.
* Attend all scheduled visits and to comply with all study procedures.
* Negative serum pregnancy test at Screening, and a negative urine pregnancy test on Day 0.

Exclusion Criteria:

* Known or suspected congenital or acquired immunodeficiency, immunosuppressive therapy such as anti-cancer chemotherapy or radiation therapy within the preceding 6 months, or long-term (at least 2 weeks within the previous 3 months) systemic corticosteroids therapy (at a dose of at least 10 mg of prednisone or equivalent), or depot preparation within the previous 3 months. Topical steroids are allowed.
* Administration of immunoglobulins and/or any blood products within 3 months before enrollment or planned administration during treatment period of study.
* Presence of acute or chronic illness associated with an oral temperature of >38.0 °C or requiring hospitalization at time of enrollment.
* Any of the following serological findings at Screening:

positive Hepatitis B surface antigen (HBsAg), positive Hepatitis C (anti-HCV), or positive human immunodeficiency virus (HIV).

* Personal or family history of thymic pathology (e.g., thymoma), thymectomy, or myasthenia.
* History of significant allergic reaction to the vaccine components
* Asplenia, functional asplenia, or any condition resulting in the absence or removal of the spleen.
* Active or potentially progressive neurologic disease or injury including but not limited to: Parkinson's, Guillain Barré, epilepsy, seizures (except febrile seizures under the age of 2), cerebrovascular accident, head trauma requiring hospitalization within the preceding 3 years, or any other neurologic condition thought to impact the integrity of the blood brain barrier.
* Clinically significant abnormal ECG findings at Screening
* Impaired hepatic function, and/or clinically significant or unexplained elevations of alanine aminotransferase (ALT, SGPT), or aspartate aminotransferase (AST, SGOT) > 3X the upper limit of normal.
* Impaired renal function, as shown by but not limited to, serum creatinine >2.0 mg/dL.
* Impaired hematopoietic function and/or clinically significant hematological laboratory abnormalities.
* A history of alcohol or drug abuse within 12 months prior to study entry.
* Pregnant or lactating women and women of childbearing potential who are not using an acceptable method of contraception at least 28 days prior to enrollment. Post menopausal women will be considered not of childbearing potential 1 year after last menstrual period.
* Behavioral, cognitive, or psychiatric disease that, in the opinion of the Investigator affects the ability of the subject to understand the scope of the study and/or unlikely to be able to be compliant with the study procedures and visits.
* Any other condition, which in the Investigator's judgment, might result in an increased risk to the subject, or would affect the subject's participation in the study.
* Participation in another clinical trial investigating a vaccine, drug or medical procedure in the 30 days preceding informed consent.
* Any vaccine administered within 30 days prior to study vaccination. Note: Influenza vaccine can be administered 1 week preceding study vaccination.
* Planned participation in another clinical trial during the present trial period.
* Planned receipt of any vaccine in the 4 weeks following the trial vaccination.
* Research site personnel or their family members cannot be enrolled as subjects in this trial.

Min Age: 50 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 479 (Actual)
Dates: Start 2008-10; Primary Completion 2009-06 (Actual); Study Completion 2009-12 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Medical Director, Study Director — Sanofi Pasteur Inc
Locations (15):
- United States (15):
  - Advanced Clinical Research Inst., Anaheim, California
  - Lynn Health Science Institute, Colorado Springs, Colorado
  - Miami Research, South Miami, Florida
  - Advanced Clinical Research- Idaho, Boise, Idaho
  - Idaho Falls Infectious diseases, Idaho Falls, Idaho
  - Johnson County Clinical Trials, Lenexa, Kansas
  - Vince & Associates, Overland Park, Kansas
  - Bio-Kinetic, Springfield, Missouri
  - Big Sky Clinical Research, Butte, Montana
  - Infectious Disease Specialists, PC, Missoula, Montana
  - Odyssey Research, Fargo, North Dakota
  - Lynn Health Science Institute, Oklahoma City, Oklahoma
  - Research Across America, Dallas, Texas
  - Benchmark, Fort Worth, Texas
  - Radiant Research, Salt Lake City, Utah

REFERENCES:
- See also: Related Info — http://www.sanofipasteur.com

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Participants were enrolled from 03 October 2008 to 08 December 2008 in 15 clinical centers in the US.
Pre-assignment Details: A total of 498 of the 479 randomized participants who met the inclusion and exclusion criteria were vaccinated. 1 subject was withdrawn from the study before receiving any study vaccine and was excluded from analysis and this report.
Groups:
- ChimeriVax WN02 Vaccine Low Dose: Participants who received ChimeriVax-WN02 vaccine at a dose of approximately 4 x 3log10 plaque forming units given one time subcutaneously
- ChimeriVax WN02 Vaccine Medium Dose: Participants who received ChimeriVax-WN02 vaccine at a dose of approximately 4 x 4log10 plaque forming units given one time subcutaneously
- ChimeriVax WN02 Vaccine High Dose: Participants who received ChimeriVax-WN02 vaccine at a dose of approximately 4 x 5log10 plaque forming units given one time subcutaneously
- Placebo: Participants who received placebo (saline) given one time subcutaneously
Period: Overall Study
Arm/Group | ChimeriVax WN02 Vaccine Low Dose | ChimeriVax WN02 Vaccine Medium Dose | ChimeriVax WN02 Vaccine High Dose | Placebo
Started | 122 | 124 | 113 | 120
Completed | 121 | 122 | 110 | 120
Not Completed | 1 | 2 | 3 | 0
Not completed — Protocol Violation | 0 | 1 | 0 | 0
Not completed — Withdrawal by Subject | 0 | 1 | 1 | 0
Not completed — Death | 0 | 0 | 2 | 0
Not completed — Participant unable to return for visit | 1 | 0 | 0 | 0

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | ChimeriVax WN02 Vaccine Low Dose | ChimeriVax WN02 Vaccine Medium Dose | ChimeriVax WN02 Vaccine High Dose | Placebo | Total
Number analyzed (Participants) | 122 | 124 | 113 | 120 | 479
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 0 | 0 | 0 | 0
  Between 18 and 65 years | 72 | 75 | 62 | 76 | 285
  >=65 years | 50 | 49 | 51 | 44 | 194
Age, Continuous [Mean (Standard Deviation); unit: Years] | 63.1 (9.39) | 62.9 (8.10) | 63.4 (9.01) | 62.2 (8.28) | 62.9 (8.69)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 76 | 65 | 63 | 64 | 268
  Male | 46 | 59 | 50 | 56 | 211
Region of Enrollment [Number; unit: Participants]
  United States | 122 | 124 | 113 | 120 | 479

OUTCOME MEASURES:

1. Primary Outcome: Geometric Mean Titers (GMTs) of Antibodies to Vaccination With ChimeriVax™ WN02 or a Placebo Vaccine
Description: Antibodies to the vaccine antigens were measured by the Plaque Reduction Neutralization Test.
Time Frame: Day 0 and Day 28 post-vaccination
Population: Serum antibody levels were assessed in the per-protocol population.
Measure: Geometric Mean (95% Confidence Interval); unit: Titers
Arm/Group | ChimeriVax WN02 Vaccine Low Dose | ChimeriVax WN02 Vaccine Medium Dose | ChimeriVax WN02 Vaccine High Dose | Placebo
Number analyzed (Participants) | 114 | 118 | 108 | 114
Titers
  Day 0 | 5.00 [5.00 to 5.00] | 5.76 [4.92 to 6.74] | 5.06 [4.94 to 5.20] | 5.22 [4.80 to 5.68]
  Day 28 | 688 [453 to 1047] | 600 [405 to 890] | 674 [464 to 978] | 5.93 [4.96 to 7.08]

2. Secondary Outcome: Number of Participants Developing Viremia After Vaccination With ChimeriVax™ WN02 or a Placebo Vaccine.
Description: Viremia is defined as number of subjects in the analysis population dose group with detected (≥ 20 Plaque forming units [pfu]/mL) viremia at the reported visit.
Time Frame: Day 2 up to Day 14 post-vaccination
Population: Viremia concentrations were assessed in a randomly selected subset of the per-protocol population.
Measure: Number; unit: Participants
Arm/Group | ChimeriVax WN02 Vaccine Low Dose | ChimeriVax WN02 Vaccine Medium Dose | ChimeriVax WN02 Vaccine High Dose | Placebo
Number analyzed (Participants) | 80 | 82 | 73 | 80
Participants
  Day 2 | 1 | 0 | 1 | 0
  Day 4 | 33 | 28 | 15 | 0
  Day 6 | 21 | 33 | 29 | 0
  Day 8 | 19 | 19 | 21 | 0
  Day 10 | 15 | 18 | 8 | 1
  Day 12 | 7 | 5 | 7 | 0
  Day 14 | 2 | 0 | 2 | 0

3. Primary Outcome: Number of Participants With Seroconversion Following Vaccination With ChimeriVax™ WN02 or a Placebo Vaccine.
Description: Antibodies to vaccine were measured by the Plaque Reduction Neutralization Test.
  Seroconversion was defined as a four-fold or greater rise in titer between pre- and post-injection samples; or a post-vaccination (Day 28) titers of ≥ 1:20 in participants with baseline titer ≤ 1:10.
Time Frame: Day 0 and Day 28 post-vaccination
Population: Serum antibody levels and seroconversion were assessed in the per-protocol population.
Measure: Number; unit: Participants
Arm/Group | ChimeriVax WN02 Vaccine Low Dose | ChimeriVax WN02 Vaccine Medium Dose | ChimeriVax WN02 Vaccine High Dose | Placebo
Number analyzed (Participants) | 114 | 118 | 108 | 114
Participants | 105 | 110 | 103 | 3

4. Primary Outcome: Number of Participants Reporting Solicited Injection Site or Systemic Reactions Following Vaccination With ChimeriVax™ WN02 or a Placebo Vaccine.
Time Frame: Day 0 up to Day 14 post-vaccination
Population: Safety assessments were on the Safety, intend-to-treat Population.
Measure: Number; unit: Participants
Arm/Group | ChimeriVax WN02 Vaccine Low Dose | ChimeriVax WN02 Vaccine Medium Dose | ChimeriVax WN02 Vaccine High Dose | Placebo
Number analyzed (Participants) | 122 | 124 | 112 | 120
Participants
  Any Pain [N = 122, 123, 112, 120] | 14 | 29 | 10 | 12
  Grade 3 Pain (Prevents daily activities) | 0 | 1 | 0 | 0
  Any Erythema [N = 122, 123, 112, 120] | 2 | 4 | 0 | 0
  Grade 3 Erythema (> 10 cm) | 0 | 0 | 0 | 0
  Any Swelling [N = 121, 123, 112, 120] | 1 | 0 | 0 | 0
  Grade 3 Swelling (> 10 cm) | 0 | 0 | 0 | 0
  Any Fever [N = 122, 123, 111, 120] | 0 | 0 | 3 | 0
  Grade 3 Fever (≥ 39.0 ºC or ≥ 102.1 ºF) | 0 | 0 | 1 | 0
  Any Headache [N = 122, 123, 112, 120] | 31 | 34 | 33 | 31
  Grade 3 Headache (prevents daily activities) | 2 | 3 | 3 | 1
  Any Malaise [N = 122, 123, 112, 120] | 26 | 26 | 27 | 25
  Grade 3 Malaise (Prevents daily activities) | 2 | 4 | 3 | 2
  Any Myalgia [N = 122, 123, 112, 120] | 28 | 25 | 22 | 20
  Grade 3 Myalgia (Prevents daily activities) | 2 | 2 | 1 | 0

ADVERSE EVENTS:
Time Frame: Adverse events data were collected from the day of vaccination (Day 0) to up to 6 months post-vaccination.
Arm/Group | ChimeriVax WN02 Vaccine Low Dose | ChimeriVax WN02 Vaccine Medium Dose | ChimeriVax WN02 Vaccine High Dose | Placebo
Serious Adverse Events (participants affected / at risk) | 4/122 | 1/124 | 3/112 | 5/120
Other Adverse Events (participants affected / at risk) | 51/122 | 56/124 | 42/112 | 54/120
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk, or affected / at risk where a term's number at risk differs (number of events):
Term (organ system) | ChimeriVax WN02 Vaccine Low Dose (N=122) | ChimeriVax WN02 Vaccine Medium Dose (N=124) | ChimeriVax WN02 Vaccine High Dose (N=112) | Placebo (N=120)
Angina pectoris (Cardiac disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Atrial fibrillation (Cardiac disorders) | 1 (1) | 0 (0) | 1 (1) | 0 (0)
Coronary artery disease (Cardiac disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Myocardial infarction (Cardiac disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Vitello intestinal duct remnant (Congenital, familial and genetic disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Influenza (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 2 (2)
Pneumonia (Infections and infestations) | 1 (1) | 0 (0) | 0 (0) | 0/0 (0)
Accidential poisoning (Injury, poisoning and procedural complications) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Subdural haematoma (Injury, poisoning and procedural complications) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Arthralgia (Musculoskeletal and connective tissue disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Benign neoplasm of thyroid gland (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Endometrial cancer stage II (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Prostate cancer metastatic (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Intracranial aneurysm (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
OTHER ADVERSE EVENTS (reported when occurring in more than 5.00% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | ChimeriVax WN02 Vaccine Low Dose (N=122) | ChimeriVax WN02 Vaccine Medium Dose (N=124) | ChimeriVax WN02 Vaccine High Dose (N=112) | Placebo (N=120)
Nasopharyngitis (Infections and infestations) | 4 (5) | 6 (6) | 6 (6) | 8 (10)
Upper respiratory tract infection (Infections and infestations) | 4 (5) | 1 (1) | 2 (2) | 8 (9)
Cough (Respiratory, thoracic and mediastinal disorders) | 7 (7) | 3 (4) | 3 (3) | 7 (8)
Injection site pain (General disorders) | 14 (14) | 29 (29) | 10 (10) | 12 (12)
Headache (Nervous system disorders) | 31 (31) | 34 (34) | 33 (33) | 31 (31)
Malaise (General disorders) | 26 (26) | 26 (26) | 27 (27) | 25 (25)
Myalgia (Musculoskeletal and connective tissue disorders) | 28 (28) | 25 (25) | 22 (22) | 20 (20)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
Sponsor must have the opportunity to review at least 60 days prior to submission for publication or presentation. If review indicates that potentially patentable subject matter would be disclosed, publication or public disclosure may be delayed for a maximum of an additional 60 days to allow for filing the necessary patent applications